CLINICAL TRIAL: NCT02619500
Title: A Pragmatically Applied Cervical and Thoracic Non-thrust Mobilizations Versus Thrust Manipulation for Patients With Mechanical Neck Pain: A Multicenter Randomized Clinical Trial
Brief Title: Thrust Manipulation vs. Non-thrust Mobilizations for Mechanical Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Youngstown State University (Other)
Collaborators: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, David W. Griswold, Assistant Professor of Physical Therapy, Youngstown State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 033-16
Record Dates: First submitted 2015-11-24; First posted 2015-12-02 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thrust Manipulation (Experimental): Subjects in this arm will receive spinal thrust manipulation to both the cervical and thoracic spines.
  Interventions: Other: Home Exercise Program; Other: Patient advice, encouragement, and education; Other: Thrust Manipulation
- Non-thrust Mobilizations (Active Comparator): Subjects in this arm will receive spinal non-thrust mobilizations to both the cervical and thoracic spines
  Interventions: Other: Home Exercise Program; Other: Patient advice, encouragement, and education; Other: Non-thrust Mobilizations

INTERVENTIONS:
Other: Home Exercise Program — A standardized home exercise program will be given to subjects that will include active range of motion of the cervical and thoracic spine and deep cervical flexion endurance exercises.
Other: Patient advice, encouragement, and education — Therapists will provide each subject with advice and education pertaining to their condition as well as encouragement towards reducing pain and disability.
Other: Thrust Manipulation — High velocity low amplitude (HVLA) thrust performed at or near the end range of a targeted segment in both the cervical and thoracic spine
  Arms: Thrust Manipulation
Other: Non-thrust Mobilizations — Repetitive and rhythmic accessory passive movements applied with either small or large amplitude at a targeted segment to both the cervical and thoracic spine
  Arms: Non-thrust Mobilizations

SUMMARY:
The purpose of this clinical trial is to compare the use of thrust manipulation to non-thrust mobilizations for mechanical neck pain when they are applied to both the cervical and thoracic spine. Both of these techniques have been compared in previous trials but a pragmatic approach will be employed as well as controlling for clinical equipoise.

DETAILED DESCRIPTION:
A total sample size of 136 subjects with mechanical neck pain will be recruited to participant in this trial from multiple clinic and university sites around the country. Each subject will be evaluated by a licensed physical therapist that specializes in orthopedic manual therapy (OMT). Each treating therapist will be blinded be the data collection and each data collection therapist will be blinded to the treatment allocation. Subjects data will be collected at the initial visit, second visit, and at discharge. The maximum number of weeks that a subject may be enrolled is 8 weeks (2 months). At that point, they are discharged from the study. The treating therapist will allocate the subject through the already completed randomization procedures. Once the subject is randomized, the treating therapist will perform the OMT based on their clinical reasoning and in a manner they feel would benefit the patient the most. In addition to the OMT, each subject will receive a home exercise program, advice, encouragement, and education. A number of outcome variables will be collected regarded pain and disability as well as one physical performance measure.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint of neck pain. (Non-specific neck pain with a primary location between the superior nuchal line and the first thoracic spinous process)
* Age >18
* A minimum Neck Disability Index (NDI) score ≥ 20%

Exclusion Criteria:

* Contraindications to OMT including; malignancy, myelopathy, fracture, metabolic disease, rheumatoid arthritis, long-term corticosteroid use.
* Nerve root compression diagnosed as having at least 2 of the following:

  * Upper extremity muscle weakness within a specific cervical/thoracic myotome
  * Diminished deep tendon reflexes of the biceps brachii, brachioradialis, or triceps muscle.
  * Diminished sensation to light touch or pinprick in a specific upper extremity dermatome.
* History of neck or thoracic spine surgery
* Neck pain of <2 on the NPRS
* Currently receiving other forms of conservative care and unwilling to stop for the duration of their participation in the study.
* Any pending litigation related to their neck pain
* Therapist is unable to elicit the chief complaint with passive accessory intervertebral movements (PAIVM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the Neck Disability Index (NDI) | 3 days and 8 weeks
  The NDI is a self-report measure of perceived disability and it is comprised of ten questions using an ordinal scale from 0 to 5 for a maximum of 50 points. The score is doubled to achieve a % score. The higher an individual scores on the NDI, the greater their perceived level of disability.

SECONDARY OUTCOMES:
Change from baseline on The Patient Specific Functional Scale (PSFS) | 3 days and 8 weeks
  The PSFS is a patient identified self-report questionnaire that measures general activity limitations. The scale ranges from 0 (unable to perform) to 10 (able to perform the activity at the level prior to injury). The patient reports three activities that are limited due to the current injury and an average rating for all three activities is calculated.
Change from baseline on The Numerical Pain Rating Scale (NPRS) | 3 days and 8 weeks
  The NPRS is an 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain). Two separate pain ratings will be collected (current and average over a 24 hour period) experienced over 24 hours and then averaged for a composite score.
Change from baseline on The Global Rating Of Change Scale (GROC) | 3 days and 8 weeks
  The GROC is a 15-point scale used to quantify a patient's improvement with treatment or to record the clinical course of a condition over time. Patients are asked to describe their overall condition since the start of treatment until the present time with options ranging from -7 ("a very great deal worse") to +7 ("a very great deal better") and 0 being described as "about the same."
Change from baseline on the Deep Cervical Flexion Endurance (DCF) | 3 days and 8 weeks
  Patients are positioned in supine and will be instructed to maximally tuck his/her chin isometrically. Patients will then be instructed to lift their head 2.5 cm off the plinth and to maintain upper cervical flexion simultaneously for as long as they were able. A skin fold along the antero-lateral neck will be monitored and the investigator's hand will remain under the occiput of the patient for tactile cueing. The timing of the position began once the patient is in the correct position and stopped if; the patient's head drops into the fingers of the clinician, is elevated greater than one inch, the patient loses the skin fold on the antero-lateral neck, or the patient is unable to continue.

OTHER OUTCOMES:
Questionnaire using a scale that rates each clinicians own Clinical Equipoise | baseline only
  Therapist equipoise will be measured globally regarding both of the orthopedic manual therapy techniques on a single scale that ranges form 0 to +2 (only a single measure. Each treating therapist will make a global opinion regarding the efficacy of non-thrust mobilization compared to thrust manipulation. An ordinal scale will be used with a score of 0 meaning that the clinician does not believe that either of the competing treatments are more beneficial than the other. The scale then ranges from +1 and +2 for both mobilizations and manipulations. The rater circles if one of the numbers depending on which of the treatments they feel are clinically more effective. See below.
  Mobilization is better Neither Manipulation is better
  +2 - 1 - 0 - +1 - +2

CONTACTS AND LOCATIONS:
Overall Officials: Josh Cleland, PhD, Study Chair — Nova Southeastern University
Locations (1):
- Youngstown state university, Youngstown, Ohio, United States

REFERENCES:
- [Background] Griswold D, Learman K, O'Halloran B, Cleland J. A preliminary study comparing the use of cervical/upper thoracic mobilization and manipulation for individuals with mechanical neck pain. J Man Manip Ther. 2015 May;23(2):75-83. doi: 10.1179/2042618614Y.0000000095. PMID 26109828
- [Background] Young JL, Walker D, Snyder S, Daly K. Thoracic manipulation versus mobilization in patients with mechanical neck pain: a systematic review. J Man Manip Ther. 2014 Aug;22(3):141-53. doi: 10.1179/2042618613Y.0000000043. PMID 25125936
- [Background] Dunning JR, Cleland JA, Waldrop MA, Arnot CF, Young IA, Turner M, Sigurdsson G. Upper cervical and upper thoracic thrust manipulation versus nonthrust mobilization in patients with mechanical neck pain: a multicenter randomized clinical trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):5-18. doi: 10.2519/jospt.2012.3894. Epub 2011 Sep 30. PMID 21979312
- [Background] Cook C, Learman K, Showalter C, Kabbaz V, O'Halloran B. Early use of thrust manipulation versus non-thrust manipulation: a randomized clinical trial. Man Ther. 2013 Jun;18(3):191-8. doi: 10.1016/j.math.2012.08.005. Epub 2012 Oct 2. PMID 23040656
- [Derived] Griswold D, Learman K, Kolber MJ, O'Halloran B, Cleland JA. Pragmatically Applied Cervical and Thoracic Nonthrust Manipulation Versus Thrust Manipulation for Patients With Mechanical Neck Pain: A Multicenter Randomized Clinical Trial. J Orthop Sports Phys Ther. 2018 Mar;48(3):137-145. doi: 10.2519/jospt.2018.7738. Epub 2018 Feb 6. PMID 29406835